CLINICAL TRIAL: NCT01835288
Title: A Phase II Study of Arsenic Trioxide in Patients With Relapsed and/or Refractory Acute Myeloid Leukemia (AML) and Mutated Nucleophosmin 1 (NPM1) Gene
Brief Title: Arsenic Trioxide in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-26938; NCI-2013-00767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMAML0023 (Other: OnCore)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (arsenic trioxide) (Experimental): Patients receive arsenic trioxide IV over 1-2 hours daily for up to 45 days. Patients achieving complete remission, receive arsenic trioxide IV over 1-2 hours daily 5 days a week for 4 weeks. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: arsenic trioxide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well arsenic trioxide works in treating patients with relapsed or refractory acute myeloid leukemia. Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the complete remission rate of relapsed and refractory acute myeloid leukemia (AML) patients with Mutated Nucleophosmin 1 (NPM1) gene.

SECONDARY OBJECTIVES:

I. Determine the duration of remission in these patients. II. Determine the in vivo biological effect of arsenic trioxide in AML with mutated NPM1.

OUTLINE:

Patients receive arsenic trioxide intravenously (IV) over 1-2 hours daily for up to 45 days. Patients achieving complete remission, receive arsenic trioxide IV over 1-2 hours daily 5 days a week for 4 weeks. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* AML, any French- American- British (FAB) subtype except M3, with confirmed mutation in the NPM1 gene
* Relapsed and/or refractory AML from any duration of complete remission (CR); any number of prior therapies allowed
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, life expectancy > 3 months
* Serum creatinine =< 2.0 mg/dL
* Bilirubin =< 2.0 mg/dL
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in women; sexually active males or females may not participate unless they have agreed to use an effective contraceptive method
* Patients who are currently receiving another investigational drug
* Patients who are currently receiving other anti-cancer agents
* Uncontrolled systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Known hypersensitivity to arsenic trioxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission following arsenic trioxide induction | After 4 weeks of therapy

SECONDARY OUTCOMES:
Median duration of remission | Time from documented complete remission until time of disease relapse, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno de Medeiros, Principal Investigator — Stanford University